CLINICAL TRIAL: NCT06146140
Title: Prospective, Double-Blinded, Randomized Placebo Controlled Study of an Oral Herbal Supplement on Photoaged Skin and Elasticity
Brief Title: Effects of an Oral Herbal Supplement on Skin Aging, Hydration, and Elasticity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Vidya Herbs (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: i23-09-Vidya_Skin_Supp
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Photoaging
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Herbal Supplement (Experimental): Oral supplement containing an herbal blend
  Interventions: Dietary Supplement: Oral herbal supplement
- Oral Placebo Supplement (Placebo Comparator): Oral placebo supplement
  Interventions: Dietary Supplement: Oral placebo supplement

INTERVENTIONS:
Dietary Supplement: Oral herbal supplement — Take one capsule daily
  Arms: Oral Herbal Supplement
Dietary Supplement: Oral placebo supplement — Take one capsule daily
  Arms: Oral Placebo Supplement

SUMMARY:
The purpose of this study is to evaluate how an oral herbal supplementation influences facial skin elasticity and facial hydration as well as markers of photoaging (erythema and pigmentation).

DETAILED DESCRIPTION:
Skin is the largest organ of the body and skin aging represents a primary indicator of the aging process in the body. Photoaging is among the most crucial factors that cause skin aging damage. Photoaged skin is primarily induced by prolonged exposure to ultraviolet radiation leading to the appearance of increased skin pigmentation, reduced elasticity, and pronounced wrinkles. There has been an increasing recognition of the influence of nutrition on skin health with dietary elements emerging as a viable alternative approach to preventing photoaging. The aim of this study is to understand how oral supplementation impacts photoaged skin, facial hydration, and facial elasticity.

ELIGIBILITY:
Inclusion Criteria:

- Women who are 35 to 55 years of age

Exclusion Criteria:

* Individuals who are pregnant or breastfeeding.
* Prisoners.
* Adults unable to consent.
* Those who are unwilling to discontinue topical probiotics, topical hydroquinone, retinoids, bakuchiol, vitamin C, or acetyl zingerone containing products for two weeks to meet the washout criteria prior to enrolling.
* Subjects with any of the following facial cosmetic treatments in the past 3 months or those who are unwilling to withhold the following facial cosmetic treatments during the study including botulinum toxin, injectable fillers, microdermabrasion, intense pulsed light (IPL), peels, laser treatments, acid treatments, facial plastic surgery, or any other medical treatment administered by a physician or skin care professional which is designed to improve the appearance of facial skin.
* Individuals who have changed any of their hormonal based contraception within 3 months prior to joining the study.
* Current tobacco smoker or a tobacco smoking history of greater than 10 pack-years.
* Any known allergy to any of the ingredients in the study product.
* Those who have been on an oral antibiotic within 1 month prior enrolling
* Those who are unwilling to discontinue oral probiotics-based supplementation or supplement ingredients found in the study's oral, product 1 month prior to enrollment

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Skin Elasticity | 8 weeks
  Skin elasticity measured with a handheld non-invasive device (Cutometer, Delfin Technologies Ltd.)
Change in Skin Hydration | 8 weeks
  The skin capacitance will be measured with a handheld non-invasive device (Skin MoistureMeterSC, Delfin Technologies Ltd.). The measurement is in arbitrary units per manufacturer.

SECONDARY OUTCOMES:
Change in skin pigmentation intensity | 8 weeks
  Facial photographs will be obtained and analyzed utilizing the BTBP 3D Clarity Pro Facial Modeling and Analysis System (Brigh-Tex BioPhotonics, San Jose, CA, USA). The measurement will analyze pigment intensity and will be reported as a relative change from baseline.
Change in appearance of facial wrinkles | 8 weeks
  Facial photographs will be obtained and analyzed utilizing the BTBP 3D Clarity Pro Facial Modeling and Analysis System (Brigh-Tex BioPhotonics, San Jose, CA, USA). The measurement will analyze wrinkle severity that is a measure of both the wrinkle depth and width and will be reported as a relative change from baseline.
Change in the skin erythema | 8 weeks
  Facial photographs will be obtained and analyzed utilizing the BTBP 3D Clarity Pro Facial Modeling and Analysis System (Brigh-Tex BioPhotonics, San Jose, CA, USA). The measurement will analyze erythema intensity and will be reported as a relative change from baseline.
Change in skin transepidermal water loss | 8 weeks
  Skin transepidermal water loss measured with a handheld non-invasive device (Vapometer, Delfin Technologies Ltd.)
Self-perception of skin (changes in facial fine lines and wrinkles, firmness, etc) | 8 weeks
  Assessed with the use of a subjective questionnaire to be completed by participants. Self-perception will be measured by rating symptoms of skin improvement, clarity, smoothness, etc.)
Product Tolerability | 8 weeks
  Assessed with the use of a tolerability questionnaire to be completed by participants. Tolerability will be measured by rating symptoms such as burning, stinging, and scaling.

IPD SHARING:
Plan to Share IPD: No